CLINICAL TRIAL: NCT01542658
Title: Comparison of Robot-assisted Laparoscopic Myomectomy With Traditional Laparoscopic Myomectomy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 100167-E
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Uterine Myoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- uterine myoma

SUMMARY:
This study is to reveal any potential advantage of Robot-assisted Laparoscopic Myomectomy (RLAM) over Traditional Laparoscopic Myomectomy (TLM) by comparing the perioperative variables and short-term outcome of RALM and TLM patients.

DETAILED DESCRIPTION:
All patients with symptomatic uterine myomas who underwent traditional laparoscopic myomectomy or robotic laparoscopic myomectomy were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* cases with uterine myoma

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uterine myoma, and underwent primary treatment (RALM and TLM) in Far Eastern Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
amount of postoperation abdominal drainage | 5 days

SECONDARY OUTCOMES:
operation time | 1 day
blood loss | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan